CLINICAL TRIAL: NCT02698891
Title: Feasibility and Safety of Avoiding Granulocyte Colony-stimulating Factor Prophylaxis During the Paclitaxel Portion of Dose Dense Doxorubicin-Cyclophosphamide and Paclitaxel Regimen
Brief Title: Avoiding Growth Factor During Paclitaxel Treatment in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nancy Lin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-516
Record Dates: First submitted 2016-03-02; First posted 2016-03-04 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Early Stage Breast Cancer
Keywords: Early Stage Breast Cancer
MeSH Terms: interventions — Paclitaxel; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel (Experimental): After the screening procedures confirm participation in the research study:
  175 mg/m^2 Paclitaxel via IV, once every 2 weeks x 4 cycles. (1 cycle = 2 weeks)
  -- Neulasta™ (Pegfilgrastim) 6 mg SQ x1 is administered on day 2 of each treatment cycle, approximately 24 hours after the chemotherapy treatment, if:
  * The patient experiences a prior episode of fever and neutropenia.
  * If the patient has an active infection this decision will be at provider discretion.
  * If Neulasta™(Pegfilgrastim) is administered in any Paclitaxel cycle for a given patient, it will be then administered for all future cycles.
  Interventions: Drug: Paclitaxel; Drug: Neulasta

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: Taxol; Onxal
Drug: Neulasta
  Other Names: Pegfilgrastim

SUMMARY:
This research study is testing the safety and feasibility of delivering the 4 cycles of 'dose-dense' paclitaxel without the use of Neulasta (Pegfilgrastim) as a Granulocyte Colony-stimulating Factor (G-CSF) support. The research study is for participants who have early stage breast cancer and have been recommended to receive a standard chemotherapy regimen, doxorubicin/cyclophosphamide (AC) plus Paclitaxel (T), in what is called a "dose-dense" fashion to prevent recurrences.

DETAILED DESCRIPTION:
Low white cell blood counts increase the risk of infections; thus, in order to give each cycle of chemotherapy, white blood cell count must have recovered adequately in between cycles. Traditionally, this regimen has been given with the use of a medicine called Neulasta (Pegfilgrastim) to speed the recovery of the white blood cell count in order to maximize the chances that the next cycle of chemotherapy can be given on time.

The names of the study interventions involved in this study are:

-- Neulasta (Pegfilgrastim)

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed Stage I-III breast cancer (as defined by the revised, American Joint Committee on Cancer 7th edition criteria) and be at sufficient risk for tumor recurrence. Staging studies to exclude metastatic disease are not required in asymptomatic patients. However, patients with findings considered suspicious for metastatic disease on any staging studies that are obtained need to be evaluated to exclude stage IV breast cancer.
* Patients must be deemed by their treating oncologist as candidates for (neo) adjuvant chemotherapy with dose dense AC and T.
* Age ≥ 18 years and < 65 at the time of informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1.
* Any grade 3 or clinically significant grade 2 treatment-related non-hematological toxicity must be resolved to grade 1 before retreatment with chemotherapy (with exception of alopecia)
* Laboratory Evaluations:

  * Adequate blood marrow function defined as:

    * Absolute neutrophil count (ANC) ≥1500 µL
    * Hemoglobin ≥9.0 g/dl
    * Platelets ≥100,000/mm3
  * Adequate hepatic function defined as:

    * Total bilirubin ≤ 1.2 institutional upper limit of normal (ULN)
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase ≤ 1.5 X upper limit normal (ULN)
  * Adequate renal function defined as:

    --- Serum creatinine ≤ 1.5 X ULN
  * Premenopausal women (including women who have had a tubal ligation and for women less than 12 months after the onset of menopause) must have a negative serum pregnancy test.
* Patients with risk factors for Hepatitis B or C should be tested (anti-hepatitis C virus (HCV) antibody, hepatitis B surface antigen [HBsAg] or Hepatitis B core antibody). Risk factors include: history of unprotected sexual intercourse, intravenous drug use, or originally from endemic regions. If infection is suspected, hepatitis B virus (HBV) DNA and HCV RNA should be requested as appropriate.
* Note: Patients with positive Hepatitis B or C serologies without known active disease must meet the eligibility requirements for ALT, AST, total bilirubin, and alkaline phosphatase and must have a normal international normalized ratio (INR) on at least two consecutive occasions, separated by at least 1 week, within the 30 day screening period.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have received previous cytotoxic chemotherapy including an AC-T regimen or previous therapeutic radiation therapy for any reason in the last 5 years. Because of possible limitations in bone marrow reserve, patients with such prior treatments are not appropriate candidates for this trial. Patients who have had prior hormonal therapy (for instance, tamoxifen for prevention of breast cancer) are eligible. Patients who have participated in a window study (treatment with an investigational agent prior to surgery for ≤2 weeks) are eligible but must have discontinued the investigational agent at least 14 days before enrollment.
* Participants who are receiving any other investigational agents
* Have had at least one prior episode of fever and neutropenia (ANC< 500/mm3 or expected to fall below < 500/mm3) during AC.
* Patients taking lithium.
* Patients receiving chronic treatment with oral steroids or another immunosuppressive agent (excluding steroids as part of the chemotherapy pre-medication or emetic medication).
* Known HIV-positive individuals or with any immunodeficiency status.
* Patients with history of hematologic disease, including myelodysplasia or bone marrow malignancies.
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to Paclitaxel, which cannot be managed by premedication.
* Currently pregnant or breast-feeding.
* Uncontrolled intercurrent illness including, not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or other significant diseases or disorders that, in the investigator's opinion, would exclude the subject from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber at Milford Regional Cancer Center, Milford, Massachusetts
  - Dana-Farber Cancer Institute at South Shore, Weymouth, Massachusetts
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaz-Luis I, Barroso-Sousa R, Di Meglio A, Hu J, Rees R, Sinclair N, Milisits L, Leone JP, Constantine M, Faggen M, Briccetti F, Block C, O'Neil K, Partridge A, Burstein H, Waks AG, Trippa L, Tolaney SM, Hassett M, Winer EP, Lin NU. Avoiding Peg-Filgrastim Prophylaxis During the Paclitaxel Portion of the Dose-Dense Doxorubicin-Cyclophosphamide and Paclitaxel Regimen: A Prospective Study. J Clin Oncol. 2020 Jul 20;38(21):2390-2397. doi: 10.1200/JCO.19.02484. Epub 2020 Apr 24. PMID 32330102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: May 2016 and November 2018
Groups:
- Paclitaxel: After the screening procedures confirm participation in the research study:
  175 mg/m^2 Paclitaxel via IV, once every 2 weeks x 4 cycles. (1 cycle = 2 weeks)
  -- Neulasta™ (Pegfilgrastim) 6 mg SQ x1 is administered on day 2 of each treatment cycle, approximately 24 hours after the chemotherapy treatment, if:
  * The patient experiences a prior episode of fever and neutropenia.
  * If the patient has an active infection this decision will be at provider discretion.
  * If Neulasta™(Pegfilgrastim) is administered in any Paclitaxel cycle for a given patient, it will be then administered for all future cycles.
  Paclitaxel
  Neulasta
Period: Overall Study
Arm/Group | Paclitaxel
Started | 127
Treated | 125
Completed | 115
Not Completed | 12
Not completed — Withdrawal by Subject | 2
Not completed — deemed ineligible | 1
Not completed — Adverse Event | 9

BASELINE CHARACTERISTICS:
Population: Baseline characteristics given for treated population.
Arm/Group | Paclitaxel
Number analyzed (Participants) | 125
Age, Continuous [Median (Full Range); unit: years] | 46 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 113
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 101
  More than one race | 0
  Unknown or Not Reported | 10
Body Surface Area [Median (Full Range); unit: m^2] | 1.81 [1.41 to 2.39]
ECOG Performance Status [Count of Participants; unit: Participants]
  0 - Fully Active | 119
  1 - Restricted | 6
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 84
  Postmenopausal | 41
Stage at Initial Diagnosis [Count of Participants; unit: Participants] — Stage I: Cancer in the breast only, or a breast cancer tumor smaller than 2 cm in diameter with lymph node cancer cell groups of 0.2mm to 2mm in diameter.
  Stage II: Cancer has either spread to the lymph nodes or is 2cm - 5cm in diameter and human epidermal growth factor receptor 2 positive.
  Stage III: Cancer may have spread to the skin or breast, or has infected 4+ axillary lymph nodes or beyond the axillary lymph nodes or near the breastbone. Another Stage II scenario is where breast tumor is 5cm in diameter or larger and there is cancer in the axillary lymph nodes of 0.2 - 2mm in diameter.
  Participants
    Stage I | 16
    Stage II | 81
    Stage III | 27
    Unknown | 1
Histology [Count of Participants; unit: Participants]
  Ductal Carcinoma | 94
  Lobular Carcinoma | 16
  Mixed Lobular and Ductal Carcinoma | 13
  Other | 2
Hormone Receptor Status [Count of Participants; unit: Participants]
  Estrogen and Progesterone Receptor Positive | 80
  Estrogen and Progesterone Receptor Negative | 44
  Unknown | 1
Chemotherapy Setting [Count of Participants; unit: Participants]
  Neoadjuvant | 57
  Adjuvant | 68

OUTCOME MEASURES:

1. Primary Outcome: Rate of Paclitaxel Treatment Completion Within 7 Weeks
Description: Rate of participants who completed Paclitaxel treatment in 7 weeks while omitting Neulasta™ (Pegfilgrastim). Neulasta is administered based on the following pre-specified safety criteria.
  * The patient experiences a prior episode of fever and neutropenia.
  * If the patient has an active infection this decision will be at provider discretion.
Time Frame: 7 Weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 125
percentage of participants | 90 [83 to 94]

2. Secondary Outcome: Rate of Grade 3-5 Neutropenia
Description: Percentage of participants experiencing grade 3-5 neutropenia per Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. while on treatment.
Time Frame: While on study, up to 6.2 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 125
percentage of participants | 8.8 [5.0 to 15.7]

3. Secondary Outcome: Rate of Grade 3-4 Toxicities, Excluding Neutropenia
Description: Percentage of participants experiencing a grade 3 or 4 toxicity excluding grade 3 or 4 neutropenia or febrile neutropenia per Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: While on study, up to 6.2 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 125
percentage of participants | 12 [7.4 to 18.9]

4. Secondary Outcome: Rate of Chemotherapy Dose Reductions
Description: Percentage of participants experiencing dose reductions due to adverse events.
Time Frame: While on treatment, up to 2.3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 125
percentage of participants | 13.6 [8.7 to 20.7]

5. Secondary Outcome: Percentage of Participants Who Received All Planned Chemotherapy Cycles
Description: Percentage of Participants who received all planned chemotherapy cycles.
Time Frame: While on treatment, up to 2.3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 125
percentage of participants | 92 [85.8 to 96.1]

6. Secondary Outcome: Rate of Hypersensitivity Reactions on Cycles 3-4 of Paclitaxel, When Steroid is Avoided
Description: The percentage of participants who experienced a hypersensitivity reaction on cycles 3 and 4 without use of dexamethasone (a steroid)..
Time Frame: While on treatment, up to 2.3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 125
percentage of participants | 2.4 [0.5 to 6.9]

7. Secondary Outcome: Number of Participants With Dose Delays by Reason for Delay
Description: Number of participants with dose delays due to various different adverse events. Adverse events classified using CTCAEv 4.0.
Time Frame: While on treatment, up to 2.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 125
Participants
  Cardiotoxicity | 1
  Febrile Neutropenia | 1
  Neutropenia without Fever | 12
  Nonhematologic Toxicity | 3
  Infection | 1
  Neurotoxicity | 3
  Other | 3

8. Secondary Outcome: Median of Savings When Omitting Pegfilgrastim From Treatment.
Description: An algorithm was used to estimated median and range of potential savings per 100 patients if the use of pegfilgrastim was omitted from treatment. The algorithm is designed assuming an average wholesale price in the United States ranging from $1,361 to $4,655 for myeloid growth factors such as filgrastim (8 days of growth factor support/cycle) and peg-filgrastim ($5,443 to $18,622 for 4 cycles on the basis of April 2019 Medicare Part B Drug Average Sales Price), and applying a 95.7% reduction in the use of pegfilgrastim during paclitaxel.
Time Frame: While on treatment, up to 2.3 months
Measure: Median (Full Range); unit: millions of dollars per 100 patients
Arm/Group | Paclitaxel
Number analyzed (Participants) | 125
millions of dollars per 100 patients | 1.1 [0.5 to 1.7]

ADVERSE EVENTS:
Time Frame: While on study, up to 6.2 months
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. Remaining AEs are classified as Other AEs (OAE). Maximum grade toxicity by type was calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term. Participants are not being evaluated based on their post-operative treatment option.
Arm/Group | Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/127
Serious Adverse Events (participants affected / at risk) | 4/127
Other Adverse Events (participants affected / at risk) | 63/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel (N=127)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Neutrophil count decreased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel (N=127)
sore spots on nails, ridging (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders ? rash to cheeks (Skin and subcutaneous tissue disorders) | 1
Ridging and sore spots (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 26
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Restrictive cardiomyopathy (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 3
Supraventricular tachycardia (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 2
Dry eye (Eye disorders) | 4
Watering eyes (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Anal pain (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 21
Oral pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 3
Edema face (General disorders) | 1
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 36
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Infusion related reaction (General disorders) | 2
Localized edema (General disorders) | 1
Pain (General disorders) | 1
Lung infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 9
CD4 lymphocytes decreased (Investigations) | 1
Creatinine increased (Investigations) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 19
Platelet count decreased (Investigations) | 3
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 4
Obesity (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 18
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Concentration impairment (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 7
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 27
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 6
Urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 19
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 7
Nail discoloration (Skin and subcutaneous tissue disorders) | 7
Nail loss (Skin and subcutaneous tissue disorders) | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 7
Hypertension (Vascular disorders) | 16
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT02698891/Prot_SAP_000.pdf